CLINICAL TRIAL: NCT07216209
Title: Exercise and the Lung Cancer Tumor Microenvironment
Brief Title: The Impact of Exercise on the Tumor Microenvironment in Patients With Lung Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00005883
Record Dates: First submitted 2024-12-10; First posted 2025-10-14 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Lung Cancer - Non Small Cell
Keywords: exercise; tumor microenvironment; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Motor Activity; Lung Neoplasms | interventions — Exercise; Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise arm (Experimental): All patients will be offered a lab exercise regimen. For completion of Aim 2, only three or four visits are necessary, amounting to approximately 4 hours of the patient's time. The initial visit will be for pre-exercise screening. If the patient is deemed healthy enough to participate, an exercise test to determine the ventilatory threshold of the participant will be conducted and the VO2 determined. In the subsequent visits, the patient will perform exercise for 30 minutes at 15% above the volunteer's ventilatory threshold. Ideally, the patients will be able to complete a minimum of three sessions prior to surgery.
  Interventions: Behavioral: EXERCISE TRAINING WITH OR WITHOUT MEDICATION

INTERVENTIONS:
Behavioral: EXERCISE TRAINING WITH OR WITHOUT MEDICATION — All patients will be offered a lab exercise regimen. For completion of Aim 2, only three or four visits are necessary, amounting to approximately 4 hours of the patient's time. The initial visit will be for pre-exercise screening. If the patient is deemed healthy enough to participate, an exercise test to determine the ventilatory threshold of the participant will be conducted and the VO2 determined. In the subsequent visits, the patient will perform exercise for 30 minutes at 15% above the volunteer's ventilatory threshold. Ideally, the patients will be able to complete a minimum of three sessions prior to surgery.

SUMMARY:
There is increased interest and knowledge about the lung cancer tumor microenvironment (TME). Investigators hypothesize that patients with better baseline physiologic health will have better post-operative outcomes and that strenuous exercise will alter the TME and genetic make-up of the tumor, improving the tumor immune response. Investigators aim to identify the peri-operative and clinical outcomes that differ based on pre-operative VO2max, HRV and resting heart rate following resection of early-stage lung cancer. The physiologic states that are individual and measurable with wearable devices include but are not limited to VO2max, heart rate variability (HRV), and average resting heart rate. Investgators hypothesize that a patient's pre-operative physiologic function with higher VO2max, HRV and lower resting heart rate will be associated with improved peri-operative and post-operative outcomes. Second, investigators will compare alterations in TME based on targeted pre-operative exercise (60-80% of their VO2 max for 75min/week x2 weeks) compared to normal activity adults following resection of early-stage lung cancer. Investigators hypothesize that strenuous exercise in the pre-operative period will impact the TME by increasing levels of cytokines.

DETAILED DESCRIPTION:
Background

Lung cancer continues to be the most common cause of cancer related death in both men and women. Patients have variable responses to treatment, whether they receive neoadjuvant therapy or surgery alone. Many of these variations can be attributed to known patient risk factors including age, smoking status, and BMI. However, there are more complex pathophysiologic factors that affect how patients respond and recover from all insults, including cancer.

Lung cancer resides in a complex milieu known as the lung tumor microenvironment (TME). The TME includes the cellular makeup of the tumor as well as factors such as IL6, PDL1 ligand, COX2, PGE2, and other cytokines. These factors can cause the TME to change in states of inflammation, such as COPD, and impact carcinogenesis (1-3). Thus, it is reasonable to assume that other physiologic alterations can change the TME. These physiologic states may be alterable and could be used to improve the efficacy of targeted therapies.

The innate and adaptive immune cells in the lung TME harbor tumor promoting and suppressing activities, which may affect clinical outcomes. Cancer associated fibroblasts (CAF) isolated from human lung cancer tissues have been shown to secrete interleukin-6 (IL-6), which then stimulates Janus kinase 2(JAK2)-signal transducers. Through this mechanism, transcription 3 (STAT3) signaling is activated and ultimately leads to increased metastasis in vivo. CAFs modulate multiple immune pathways in the TME, as they also express PDL1 to blunt activation of T cells and cross present antigens to eliminate antigen-specific CD8+T cells via PDL2 and FASL. CAFs have been found to be indicators of poor prognosis, associated with nodal metastases and increased risk of recurrence (6).

Physical fitness and moderate intensity exercise training have been shown to improve immune responses to vaccination, reduce chronic low-grade inflammation, and improve various immune markers in several disease states including cancer, HIV, cardiovascular disease, diabetes, cognitive impairment, and obesity (4). In mouse models, exercise has been shown to decrease tumor incidence and growth by over 60% (5). Prior work by Simpson and colleagues have shown that even a single bout of aerobic exercise greatly increases NK cell and γδ T cell numbers as well as increases the proportion of total lymphocytes found in the peripheral blood. Exercise can also increase the number of cytotoxic T cells in the blood without increasing their proportion of total lymphocytes.

This study will capture the baseline physiologic state of patients with resectable lung cancer pre-operatively. The parameters captured will include but are not limited to: VO2max, heart rate variability (HRV), and average resting heart rate. Next, investigators will perform strenuous exercise on a subset of these patients and correlate this data with their TME and clinical peri-operative and post-operative outcomes. The TME will be evaluated with flow cytometry and real-time PCR after tumor resection and levels of IL1b, 4,6,11,12, TNFa, MCP1, TGFb, CD4 and 8 will be identified as well as the presence of PDL-1, EGFR mutations, ALK, ROS1, KRAS, BRAF.

In our clinical pilot data, strenuous exercise patients had important trends. Patients who self-reported strenuous exercise had better lung function, shorter time from diagnosis to surgery, more left sided tumors, shorter hospital LOS, and less prolonged air leaks. Long term outcomes are still pending regarding recurrence and overall survival.

Investigators hypothesize that patients with better baseline physiologic health will have better post-operative outcomes and that strenuous exercise will alter the TME and genetic make-up of the tumor, improving the tumor immune response to targeted therapies.

Specific Aims

Aim 1: Identify the peri-operative and clinical outcomes that differ based on pre-operative VO2max, HRV and resting heart rate following resection of early-stage lung cancer. The physiologic states that are individual and measurable with wearable devices include but are not limited to VO2max, heart rate variability (HRV), and average resting heart rate. Investigators hypothesize that a patient's pre-operative physiologic function with higher VO2max, HRV and lower resting heart rate will be associated with improved peri-operative and post-operative outcomes.

Aim 2: Compare alterations in TME based on targeted pre-operative exercise (60-80% of their VO2 max for 75min/week x2 weeks) compared to normal activity adults following resection of early-stage lung cancer. Investigators hypothesize that strenuous exercise in the pre-operative period will impact the TME by increasing levels of cytokines.

Significance

There is increased interest and knowledge about the lung cancer TME. There are data that demonstrate that alterations in the TME can occur based on inflammation. The literature also shows that increased level of CD8 and PDL1 expression are associated with better response to anti-PD-1 treatment (7). This occurs through the binding of PD-L1 to its receptors, which suppresses T-cell migration, proliferation and secretion of cytotoxic mediators and restricts tumor cell killing.. The PD-L1-PD-1 axis protects the host from overactive T-effector cells not only in cancer but also during microbial infections (8). If investigators can alter the level of cytokines and PD-LI expression with strenuous exercise, then patients: 1) may have improved operative outcomes, 2) could experience altered (improved) TME and may demonstrate improved response to targeted therapies.

Research Plan

Patients will be recruited from three busy thoracic surgery clinics, which see at least 30 lung cancer patients per month. All patients will be given a wearable device to record their physiologic data 24 hours/day for 2-3 weeks pre-operatively. This data will include VO2 max, HRV, resting heart rate and sleep score. The patients' peri-operative and post-operative outcomes will be recorded in a database and this data will then be linked to the patients' recorded physiologic data.

In addition to this baseline monitoring, all patients will be offered a lab exercise regimen. For completion of Aim 2, only three or four visits are necessary, amounting to approximately 4 hours of the patient's time. The initial visit will be for pre-exercise screening. If the patient is deemed healthy enough to participate, an exercise test to determine the ventilatory threshold of the participant will be conducted and the VO2 determined. In the subsequent visits, the patient will perform exercise for 30 minutes at 15% above the volunteer's ventilatory threshold. Ideally, the patients will be able to complete a minimum of three sessions prior to surgery. Those who are not able to participate due to interest or limitations in travel or physical limitations will serve as the control group.

Lung cancer specimens will be collected from all patients at the time of surgery. Investigators will perform flow cytometry and real-time PCR to identify levels of IL1b, 4,6,11,12, TNFa, MCP1, TGFb, CD4 and 8, and the presence of PDL-1, EGFR mutations, ALK, ROS1, KRAS, BRAF.

The next steps for this study will be to reproduce these experiments in a mouse model that has been previously performed by the collaborating lab. In this model investigators will be able to give targeted therapies, such as, PDL-1 inhibitors and measure the rate of response with and without strenuous exercise.

ELIGIBILITY:
Inclusion Criteria:

* lung cancer
* low risk for submaximal exercise testing in accordance with the risk stratification guidelines published by the American Heart Association and the American College of Sports Medicine (AHA/ACSM criteria).

Exclusion Criteria:

* younger than 18 years of age
* select a condition on the ACSM-AHA pre-exercise screening questionnaire indicating that physician approval is required prior to exercise
* body mass index of >30 kg/m2
* waist girth of >102cm for men and >88cm for women
* have chronic/debilitating arthritis
* have been bedridden in the past three months
* have common illness (i.e. colds) within the past 6-weeks
* HIV
* hepatitis
* history of stroke
* major affective disorder
* autoimmune disease
* pregnancy or are breast-feeding
* history of severe anaphylactic reaction to an allergen
* present with more than one of the following CVD risk factors: family history of myocardial infarction, coronary revascularization, or sudden death before 55 years of age in father or other male first-degree relative or before 65 years of age in mother or other female first-degree relative

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2030-01-15 (Estimated); Study Completion 2030-01-15 (Estimated)

PRIMARY OUTCOMES:
Tumor Microenvironment | Baseline, Perioperative, up to 24 months
  Lung cancer specimens will be collected from all patients at the time of surgery. Investigators will perform real-time PCR to identify levels of PDL-1

SECONDARY OUTCOMES:
Recurrence and Survival | Baseline, Perioperative, up to 24 months
  Patients will be compared for evidence of recurrence and followed for long-term survival

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Worrell, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
This is a local study and there are no plans to share individual patient data with outside researchers at this time.

REFERENCES:
- [Background] Tan Z, Xue H, Sun Y, Zhang C, Song Y, Qi Y. The Role of Tumor Inflammatory Microenvironment in Lung Cancer. Front Pharmacol. 2021 May 17;12:688625. doi: 10.3389/fphar.2021.688625. eCollection 2021. PMID 34079469
- [Background] Ito M, Ishii G, Nagai K, Maeda R, Nakano Y, Ochiai A. Prognostic impact of cancer-associated stromal cells in patients with stage I lung adenocarcinoma. Chest. 2012 Jul;142(1):151-158. doi: 10.1378/chest.11-2458. PMID 22302300
- [Background] Herbst RS, Soria JC, Kowanetz M, Fine GD, Hamid O, Gordon MS, Sosman JA, McDermott DF, Powderly JD, Gettinger SN, Kohrt HE, Horn L, Lawrence DP, Rost S, Leabman M, Xiao Y, Mokatrin A, Koeppen H, Hegde PS, Mellman I, Chen DS, Hodi FS. Predictive correlates of response to the anti-PD-L1 antibody MPDL3280A in cancer patients. Nature. 2014 Nov 27;515(7528):563-7. doi: 10.1038/nature14011. PMID 25428504
- [Background] Zhang L, Chen Y, Wang H, Xu Z, Wang Y, Li S, Liu J, Chen Y, Luo H, Wu L, Yang Y, Zhang H, Peng H. Massive PD-L1 and CD8 double positive TILs characterize an immunosuppressive microenvironment with high mutational burden in lung cancer. J Immunother Cancer. 2021 Jun;9(6):e002356. doi: 10.1136/jitc-2021-002356. PMID 34140315
- [Background] Rosero ID, Ramirez-Velez R, Lucia A, Martinez-Velilla N, Santos-Lozano A, Valenzuela PL, Morilla I, Izquierdo M. Systematic Review and Meta-Analysis of Randomized, Controlled Trials on Preoperative Physical Exercise Interventions in Patients with Non-Small-Cell Lung Cancer. Cancers (Basel). 2019 Jul 5;11(7):944. doi: 10.3390/cancers11070944. PMID 31284372
- [Background] Simpson RJ, Campbell JP, Gleeson M, Kruger K, Nieman DC, Pyne DB, Turner JE, Walsh NP. Can exercise affect immune function to increase susceptibility to infection? Exerc Immunol Rev. 2020;26:8-22. PMID 32139352
- [Background] Puchelle E, Zahm JM, Tournier JM, Coraux C. Airway epithelial repair, regeneration, and remodeling after injury in chronic obstructive pulmonary disease. Proc Am Thorac Soc. 2006 Nov;3(8):726-33. doi: 10.1513/pats.200605-126SF. PMID 17065381
- [Background] Wang J, Linxweiler M, Yang W, Chan TA, Morris LGT. Immunomodulatory and immunotherapeutic implications of tobacco smoking in squamous cell carcinomas and normal airway epithelium. Oncotarget. 2019 Jun 11;10(39):3835-3839. doi: 10.18632/oncotarget.26982. eCollection 2019 Jun 11. PMID 31231463